CLINICAL TRIAL: NCT05517720
Title: An Exploratory Investigation of a Novel Skincare Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trophy Skin (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20245
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Wrinkle; Photoaging; Acne; Skin Inflammation
Keywords: wrinkles; fine lines; photoaging; sun spots; acne; enlarged pores; skin health
MeSH Terms: conditions — Acne Vulgaris; Dermatitis; Melanosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aria Trio complete Facial System (Experimental): Skincare system targetting wrinkles, pore size, sun spots, and overall skin quality.
  Interventions: Other: Aria Trio complete Facial System

INTERVENTIONS:
Other: Aria Trio complete Facial System — Renew Serum, Brighten Serum, and Refine Serum.

SUMMARY:
This trial will assess the effectiveness of the Aria Trio Complete Facial system in being able to reduce blemishes, lines, and wrinkles. This skincare system that has three different functions in association with three unique serums. It is hypothesized that this customized skincare system will improve skin quality, reduce wrinkles, and reduce other skin related issues.

ELIGIBILITY:
Inclusion Criteria:

* Must experience early-stage wrinkles that are not treated by topical or oral prescription drugs/medication
* Must experience early-stage wrinkles that are not treated by over the counter products (e.g. Adapalene/Differin)
* May experience hyperpigmentation and/or dark spots
* In good general health
* Willing to follow the study protocol skincare routine
* Willing and able to share feedback and take skin pictures via the technology portal
* Discontinue use of any alpha-hydroxy acids (AHAs) or over the counter exfoliating, polishing, or peeling topical skincare treatments 1 week before and for the duration of the study.

Exclusion Criteria:

* Anyone with a diagnosed skin condition on their face
* Use of prescription medication relevant to the skin
* Undergoing any cosmetic procedures during the study including Botox, laser, or chemical peel treatments
* Use of oral acne treatment (e.g., Accutane)
* Severe chronic conditions, including oncological conditions or psychiatric disorders.
* Is pregnant, attempting pregnancy, or breastfeeding

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of the Aria Trio Complete Facial System in being able to reduce blemishes, lines, and wrinkles. | 4 weeks
  Blemishes, lines, and wrinkles will be examined using photos taken by the participants at three timepoints during the study.

SECONDARY OUTCOMES:
To determine the effectiveness of the Aria Trio Complete Facial System being able to improve perceptions of wrinkles, pore size, sun spots, and overall skin quality | 4 weeks
  Participants will be given surveys at three timepoints so that they can assess the effectiveness of the product over the 4-week trial period

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, PhD, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided